CLINICAL TRIAL: NCT05795036
Title: Using a mHealth Intervention to Promote Physical Activity in Phase III Cardiac Rehabilitation Clients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth University (Other)
Responsible Party: Principal Investigator, Chia-Wei Fan, Investigator, AdventHealth University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1848850-2
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Cardiac Rehabilitation; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Masking Description: Participants will be randomly assigned to either the intervention group or the control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Hope Clinic (Experimental): Participants will be recruited from clients admitted to the Phase III CR program at Hope Clinic. An information sheet introducing this study will be provided to clients by the assigned therapist at the Hope clinic after admission.
  Interventions: Device: mHealth 1; Device: mHealth 2

INTERVENTIONS:
Device: mHealth 1 — Participants will use Fitbit device to self-monitor their physical activity in 8 weeks.
Device: mHealth 2 — Participants will use Fitbit device to self-monitor their physical activity in 8 weeks. In addition, they will receive daily motivational text message.

SUMMARY:
In this study, the investigators will implement a pilot project of using activity tracker (i.e., Fitbit) with phase III CR clients. The study will record the participants' daily steps and sleep patterns for 8 consecutive weeks in natural settings. Two specific aims are identified for this project:

1. Develop an intervention protocol using mHealth to promote Phase III CR clients' self-monitoring of PA.
2. Examine the efficacy of the intervention on clients' PA, sleep patterns, functional capacity and QoL.

DETAILED DESCRIPTION:
In this study, the investigators will implement a pilot project of using activity tracker (i.e., Fitbit) with phase III CR clients. The study will record the clients' daily steps and sleep patterns for 8 consecutive weeks in natural settings. Two specific aims are identified for this project:

1. Develop an intervention protocol using mHealth to promote Phase III CR clients' self-monitoring of PA.
2. Examine the efficacy of the intervention on clients' PA, sleep patterns, functional capacity and QoL.

ELIGIBILITY:
Inclusion Criteria:

* currently receiving Phase III CR at Hope Clinic
* are 18 years of age or older
* can read and communicate in English
* able to follow instructions to walk
* provided signed informed consent
* willing to wear Fitbit throughout the study
* owns a smartphone with text messaging capability (participants need to decide ahead of time if they have a phone plan that is compatible with taking additional text messages without undue financial burden for themselves)
* willing to receive text messages and phone calls from the research team.

Exclusion Criteria:

* are pregnant or lactating
* have scheduled surgery or traveling within the next 8 weeks
* currently participating in other health promotion program
* sufficiently or overly active, as determined by a physical activity monitor worn for one week, indicating averaging ≥ 7,500 steps per day ("somewhat overly active").

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-02-17 (Actual); Primary Completion 2025-08-17 (Estimated); Study Completion 2025-12-17 (Estimated)

PRIMARY OUTCOMES:
Clients' demographic information will be obtained using a paper questionnaire administered at screening phase | 12 months
  Descriptive statistics will be used to assess completeness of study data, normality of outcome measures, and potential covariates, and to identify potential covariate imbalances between study arms

CONTACTS AND LOCATIONS:
Locations (1):
- AdventHealth University, Orlando, Florida, United States